CLINICAL TRIAL: NCT03288870
Title: International Multi-center Open-label Randomized Clinical Trial of Efficacy, Safety and Pharmacokinetics of BCD-100 (JSC "BIOCAD", Russia) Monotherapy Compared to Docetaxel as Second-line Therapy of Patients With Advanced Inoperable or Metastatic Non-small Cell Lung Cancer
Brief Title: Efficacy, Safety and Pharmacokinetics of BCD-100 (Anti-PD-1) Monotherapy as Second Line Treatment in Patients With Non-Small Cell Lung Cancer (DOMINUS)
Acronym: DOMINUS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-100-2/DOMINUS
Record Dates: First submitted 2017-08-23; First posted 2017-09-20 (Actual); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Non Small Cell Lung Cancer Stage IIIB; Non-Small Cell Carcinoma of Lung, TNM Stage 4
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BCD-100 monotherapy (Experimental): Patients will receive solution of BCD-100 in a dose 3 mg/kg every 3 weeks as intravenous infusion until progression of the disease or signs of intolerable toxicity
  Interventions: Drug: BCD-100
- Docetaxel monotherapy (Active Comparator): Patients will receive solution of docetaxel in a dose 75 mg per square meter every 3 weeks as intravenous infusion until progression of the disease or signs of intolerable toxicity, maximum 6 cycles
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: BCD-100 — monoclonal antibody to PD-1 receptor
  Arms: BCD-100 monotherapy
Drug: Docetaxel — Chemotherapy drug (taxane)
  Arms: Docetaxel monotherapy

SUMMARY:
International multi-center open-label randomized clinical trial of efficacy, safety and pharmacokinetics of BCD-100 (JSC BIOCAD, Russia) monotherapy compared to docetaxel as second-line therapy of patients with advanced inoperable or metastatic non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

* Verified diagnosis of non-small cell lung cancer
* Verified progression of the disease after or during first-line chemotherapy based on platinum drugs
* Absence of mutation of EGFR and ALK genes
* ECOG score 0-1
* At least one lesion, that is measurable according to RECIST 1.1 criteria
* Absence of severe organ pathology
* Anticipated live duration more that 12 weeks after screening
* Brain metastases with clinical symptoms requiring glucocorticoids and/or anticonvulsant drugs

Exclusion Criteria:

* EGFR and/or ALK mutations
* Patients with severe of live-threatening acute complications of the disease
* Intersticial lung diseases or pneumonitis
* Concomitant diseases that affect safety evaluation
* Autoimmune diseases
* Endocrine diseases that could not be compensated by hormonal therapy
* Patient needs glucocorticoids
* Significant liver or renal diseases
* Lactate dehydrogenase exceeds upper limit of normal more that 2-fold
* More that 1 chemotherapy lines for advanced/metastatic non-small cell lung cancer treatment
* Anti-tumor treatment ending less then 28 days before screening
* Prior therapy with anti-CTLA4 and/or anti-PD-1/PD-L1/PD-L2 drugs
* Prior therapy with docetaxel
* Concomitant oncological diseases except treated cervical carcinoma in situ or radically resected squamous-cell carcinoma
* Allergy to drugs based on monoclonal antibodies or docetaxel or polysorbate 80, severe reactions to paclitaxel
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2017-09-19 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2021-08-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 year
  Percent of patients who are alive after 1 year of therapy

SECONDARY OUTCOMES:
Overall response rate | 1 year
  Percent of patients who have complete or partial response to therapy
Progression-free survival | 1 year
  Percent of patients who are alive after 1 year of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Roman A Ivanov, PhD, Study Director — Vice President R&D, JSC BIOCAD
Locations (8):
- Gomel Regional Clinical Oncology Dispensary, Homyel, Belarus
- Russia (7):
  - Arkhangelsk District Clinical Oncology Dispensary, Arkhangelsk
  - Clinical Oncology Dispensary N1, Krasnodar
  - N.N. Burdenko General Military Clinical Hospital, Moscow
  - Pyatigorsk Oncology Center, Pyatigorsk
  - Saint Petersburg City Clinical Oncology Center, Saint Petersburg
  - N.N.Petrov Oncology Research Center, Saint Petersburg
  - Republican Clinical Oncology Dispensary of Ministry of Health republic Bashkortostan, Ufa

IPD SHARING:
Plan to Share IPD: No